CLINICAL TRIAL: NCT01071044
Title: Use of Lisdexamfetamine Dimesylate in Treatment of Cognitive Impairment (Chronic Fatigue Syndrome): A Double Blind, Placebo Controlled Study
Brief Title: Efficacy and Safety of Lisdexamfetamine Dimesylate in Adults With Chronic Fatigue Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rochester Center for Behavioral Medicine (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Joel L. Young, M.D., Principal Investigator, Rochester Center for Behavioral Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCBM11
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Chronic Fatigue Syndrome; Cognitive Impairments
Keywords: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Cognitive Dysfunction | interventions — Lisdexamfetamine Dimesylate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisdexamfetamine Dimesylate (Active Comparator): Subjects will be started with a single pill containing 30mg of LDX or comparable placebo, depending on the treatment assignment. At the week 2 visit, the dose will be increased to 50 mg (or comparable placebo) if the patient exhibits no significant adverse effects as judged by the Investigator. At the week 4 visit, the dose will be increased to 70 mg (or comparable placebo) if the patient exhibits no significant adverse effects as judged by the investigator.
  Interventions: Drug: Lisdexamfetamine Dimesylate
- Sugar pill (Placebo Comparator): Matching Placebo "30, 50 or 70 mg"
  Interventions: Drug: Placebo "30, 50 or 70 mg"

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate — Will be randomly assigned to one of two treatment arms in a 1:1 ratio of either LDX or placebo for 6 weeks. Subjects will be started with a single pill containing 30mg of LDX or comparable placebo, depending on the treatment assignment. At the week 2 visit, the dose will be increased to 50 mg (or comparable placebo) if the patient exhibits no significant adverse effects as judged by the Investigator. At the week 4 visit, the dose will be increased to 70 mg (or comparable placebo) if the patient exhibits no significant adverse effects as judged by the investigator.
  Other Names: Vyvanse
  Arms: Lisdexamfetamine Dimesylate
Drug: Placebo "30, 50 or 70 mg" — Will be randomly assigned to one of two treatment arms in a 1:1 ratio of either LDX or placebo for 6 weeks. Subjects will be started with a single pill containing 30mg of LDX or comparable placebo, depending on the treatment assignment. At the week 2 visit, the dose will be increased to 50 mg (or comparable placebo) if the patient exhibits no significant adverse effects as judged by the Investigator. At the week 4 visit, the dose will be increased to 70 mg (or comparable placebo) if the patient exhibits no significant adverse effects as judged by the investigator.
  Other Names: Sugar pill
  Arms: Sugar pill

SUMMARY:
Over the past decade, the Rochester Center for Behavioral Medicine (RCBM) has evaluated many patients with attention deficit hyperactivity disorder (ADHD). A recurrent finding in these patients is a history of unexplained fatigue and musculoskeletal pain.

Treatment of these patients in our clinic has revealed that when their underlying ADHD is treated with psychostimulant medication, many patients report significant improvements with regard to their fatigue and musculoskeletal pain. Patients report less subjective fatigue and pain and note overall functional improvement, although the initial and primary objective was the treatment of their attention or hyperactivity problems. We speculate that stimulants are efficacious by offering two distinct clinical properties. 1) anti-fatigue properties and 2) properties that allow patients to filter out extraneous stimuli (i.e. chronic muscle pain).

DETAILED DESCRIPTION:
As a result of these findings RCBM developed a chronic fatigue/fibromyalgia clinic in the early 2000's. This clinic was staffed by a board-certified rheumatologist and the psychiatric staff at RCBM. Through the major referral hospital in the area, patients with self-identified fibromyalgia and chronic fatigue were referred to our clinic. Over eighteen months, we evaluated 75 patients, and found that in patients who had comprehensive evaluations, nearly 70 percent also had a history of ADHD, inattentive or combined types. Diagnosis was made using clinical history and standardized symptom checklists. Oftentimes, the ADHD had been previously undiagnosed. This finding supports the link between ADHD and FMS/CFS.

Results from these evaluations reinforced our initial findings: patients who are treated for their ADHD symptoms also show a reduction in their chronic pain and fatigue symptoms. This is true regardless of previous (unsuccessful) therapies to treat their fibromyalgia.

As a result of these findings, we are conducting a controlled study to further demonstrate the efficacy of lisdexamfetamine dimesylate (LDX) in controlling fatigue symptoms in patients presenting with chronic fatigue syndrome. This is a double-blind, placebo-controlled study over a period of 8 weeks, where subjects are randomized to either LDX or placebo. We will evaluate subjects through standardized pain, fatigue and ADHD assessment scales.

ELIGIBILITY:
Inclusion Criteria:

* BRIEF-A Global Executive Composite score (GEC) ≥ 65, or Behavioral Regulation Index score (BRI) ≥ 65, or Metacognition Index score (MI) ≥ 65.
* Subjects must meet consensus criteria for chronic fatigue syndrome.
* Provide written informed consent for participation in the trial before completing any study-related procedures.
* 18-60 years at time of consent
* Male or non-pregnant females who are not breastfeeding.
* Females of reproductive potential must agree to use a medically accepted means of contraception when engaging in sexual intercourse at any time during the study.
* Are able to swallow study medication.

Exclusion Criteria:

* CFS and executive functioning impairment are not present or not diagnosable
* Serious comorbid psychiatric condition
* Subjects who were pregnant, nursing, or intended to become pregnant
* Subjects who had been on a psychostimulant regimen in the last six months
* Subjects who had a medical condition that would have been affected by psychostimulant medication
* Subjects who were of low intelligence, or who were unable to communicate effectively with the study team

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel L. Young, M.D., Principal Investigator — Rochester Center for Behavioral Medicine
Locations (1):
- Rochester Center for Behavioral Medicine, Rochester Hills, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study site began recruiting for the trial in Oct 2009 and the last subject completed the final visit on 3/7/11. Recruitment was done from within the Rochester Center (a private mental health practice), as well as some local advertising and community outreach.
Groups:
- Lisdexamfetamine Dimesylate: Subjects will be started with a single pill containing 30mg of LDX or comparable placebo, depending on the treatment assignment. At the week 2 visit, the dose will be increased to 50 mg (or comparable placebo) if the patient exhibits no significant adverse effects as judged by the Investigator. At the week 4 visit, the dose will be increased to 70 mg (or comparable placebo) if the patient exhibits no significant adverse effects as judged by the investigator.
  Lisdexamfetamine Dimesylate : Will be randomly assigned to one of two treatment arms in a 1:1 ratio of either LDX or placebo for 6 weeks. Subjects will be started with a single pill containing 30mg of LDX or comparable placebo, depending on the treatment assignment. At the week 2 visit, the dose will be increased to 50 mg (or comparable placebo) if the patient exhibits no significant adverse effects as judged by the Investigator. At the week 4 visit, the dose will be increased to 70 mg (or comparable placebo).
- Sugar Pill: Placebo Comparator: Sugar pill : Will be randomly assigned to one of two treatment arms in a 1:1 ratio of either LDX or placebo for 6 weeks. Subjects will be started with a single pill containing 30mg of LDX or comparable placebo, depending on the treatment assignment. At the week 2 visit, the dose will be increased to 50 mg (or comparable placebo) if the patient exhibits no significant adverse effects as judged by the Investigator. At the week 4 visit, the dose will be increased to 70 mg (or comparable placebo) if the patient exhibits no significant adverse effects as judged by the investigator.
Period: Overall Study
Arm/Group | Lisdexamfetamine Dimesylate | Sugar Pill
Started | 15 | 11
Completed | 13 | 11
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisdexamfetamine Dimesylate | Sugar Pill | Total
Number analyzed (Participants) | 15 | 11 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 11 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in BRIEF-A
Description: The BRIEF-A (Behavior Rating Inventory of Executive Function-- Adult Form) is comprised of the following sub-scales: Metacognition Index, Behavioral Regulation Index, Inhibit, Shift, Emotional Control, Self-Monitor, Initiate, Working Memory, Plan/Organize, Task Monitor, and Organziation of Material. These subscales are summed to provide the GEC or Global Executive Composite. Listed below are the mean improvement scores on the GEC index from baseline to endpoint. The Global Executive Composite raw score range is 70-182, with higher scores indicating more compromised executive functioning. The scores listed in the table depict mean improvement on the GEC from the beginning to the end of the study.
Time Frame: Baseline and end of study (6 weeks), assessed every 2 weeks with last observation carried forward
Population: All participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Treatment Group: Lisdexamfetamine Dimesylate 30, 50 or 70 mg
- Control Group: Placebo "30, 50 or 70 mg"
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 15 | 11
Scores on a scale | 21.38 (15.85) | 3.36 (7.26)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; These scores were calculated by subtracting participants' endpoint scores from their initial baseline scores. These change scores show the total change in executive functioning over the course of the trial. Higher values indicate improved executive functioning at the end of the trial compared to the beginning; Test type: Superiority or Other; p = .005, ANOVA; These data were initially analyzed with a one-way ANOVA

2. Secondary Outcome: Change in Fatigue Severity Scale (FSS)
Description: The Fatigue Severity Scale is designed to measure the impact of fatigue on the life of the subject. It is a nine-question likert scale survey with a raw score range of 0-63. Scores of 36 and above indicate significant fatigue. In this study, we compared the mean change in the Fatigue Severity Scale (FSS) from baseline to endpoint between LDX and placebo treated patients.
Time Frame: Baseline and end of study (6 weeks), assessed every 2 weeks with last observation carried forward
Population: All participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 15 | 11
Scores on a scale | 20.92 (14.71) | 5.00 (11.73)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.008, ANOVA

3. Secondary Outcome: Change in Hamiliton Anxiety Inventory
Description: The Hamilton Anxiety Scale is a 14-items clinician-rated scale designed to measure anxiety severity. Each of the 14 items is scored from 0 (symptom not persent) to 4 (severe symptom). The total range is 0-56. A total score of less than 17 indicates mild severity, 18-24 indicates mild to moderate severity, and a score of 25-30 indicates moderate to severe symptoms. In this study, we compared the mean change in the Hamilton Anxiety scale from baseline to week 6 between LDX and placebo-treated patients.
Time Frame: Baseline and end of study (6 weeks), assessed every 2 weeks with last observation carried forward
Population: All participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 15 | 11
Scores on a scale | 11.31 (9.74) | 6.18 (8.28)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.183, ANOVA

4. Secondary Outcome: Change in Short Form McGill Pain Questionnaire
Description: The McGill Pain Questionniare (Short Form) consists of 15 pain descriptors (11 sensory; 4 affective) which are rated on an intensity scale. 0 = none, 1 = mild, 2 = moderate or 3 = severe. The sum of the intensity scores of the words chosen for sensory, affective and total descriptors are added for a total score. The score range is 0-45. In this study, we compared the change in the Short Form McGill Pain Questionnaire (SF-MPQ) from baseline to week 6 between LDX and placebo treated patients.
Time Frame: Baseline and end of study (6 weeks), assessed every 2 weeks with last observation carried forward
Population: All participants were included in analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Lisdexamfetamine Dimesylate: Lisdexamfetamine Dimesylate 30, 50, 70 mg
- Control Group: Placebo "30, 50, or 70mg"
Arm/Group | Lisdexamfetamine Dimesylate | Control Group
Number analyzed (Participants) | 15 | 11
Scores on a scale | 10.38 (8.84) | 2.45 (9.53)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.046, ANOVA

5. Secondary Outcome: Change in Fibromyalgia Impact Questionnaire (FIQ)
Description: The Fibromyalgia Impact Questionnaire (FIQ) is an assessment that quantifies the impact of fibromyalgia on an individual, including questions on pain level, fatigue, sleep disturbance, and psychological distress, among others. The score range is 0 to 100, with higher number indicating higher Fibromyalgia severity/impact.
  Below, we compare the mean change in the Fibromyalgia Impact Questionnaire (FIQ) from baseline to week 6 between LDX and placebo treated patients.
Time Frame: Baseline and end of study (6 weeks), assessed every 2 weeks with last observation carried forward
Population: All participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 15 | 11
Scores on a scale | 20.90 (25.54) | 8.83 (18.14)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.219, ANOVA

6. Secondary Outcome: Change in Attention-Deficit Hyperactivity Disorder Rating Scale (ADHD-RS)
Description: The Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) is an 18-item scale based on DSM-IV criteria for ADHD. Each item is rated using a likert scale from 0 (none) to 3 (severe), with a total score range of 0-54, with higher scores indicating more symptoms/severity. In this study, we compared mean change in ADHD-RS total score from baseline to endpoint of the study.
Time Frame: Baseline and end of study (6 weeks), assessed every 2 weeks with last observation carried forward
Population: All participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Treatment Group: Lisdexamfetamine Dimesylate, 30, 50 or 70 mg
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 15 | 11
Scores on a scale | 18.17 (11.95) | 8.73 (7.80)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.038, ANOVA

7. Secondary Outcome: Change in Clinical Global Impression (Severity)
Description: The Clinical Global Impression (Severity) is a one-item, 7-point clinician-rated scale to assess severity of subject's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). The clinician rates the subject based on perceived severity of psychopathology, with higher numbers indicating higher severity. In this study, we compared the mean change in severity from baseline to endpoint.
Time Frame: Baseline and end of study (6 weeks), assessed every 2 weeks with last observation carried forward
Population: All participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 15 | 11
Scores on a scale | 1.92 (1.50) | .64 (.92)
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.022, ANOVA

ADVERSE EVENTS:
Time Frame: Each subject had a period of 10 weeks at which they could report any adverse events.
Groups:
- Treatment Group: Lisdexamfetamine Dimesylate 30, 50, or 70 mg
Arm/Group | Treatment Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/11
Other Adverse Events (participants affected / at risk) | 8/15 | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than .04% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=15) | Control Group (N=11)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decreased Appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry Mouth (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Facial Tics (Nervous system disorders) | 1 (1) | 0 (0)
Headaches (Nervous system disorders) | 4 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sinus Infection (Ear and labyrinth disorders) | 0 (0) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Weight Loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Relatively small sample size, imbalance of participants in active vs. placebo group due to pre-randomization, heterogenous sample (only one male participant in the study, who was in the control group and not the treatment group).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No